CLINICAL TRIAL: NCT06346535
Title: PrimeCog: Cognitive Profile, Psychosocial Characteristics, Brain MRI and Biomarkers for Stress and Neurodegeneration in Patients With Depression or Stress Induced Exhaustion Disorder in Primary Care.
Brief Title: PrimeCog: Primary Care Cognitive Testing
Acronym: PrimeCog
Status: Recruiting | Type: Observational
Sponsor: Region Östergötland (Other)
Responsible Party: Principal Investigator, Hanna Israelsson Larsen, Principal Investigator, Region Östergötland
Other Study IDs: 2022-05703-01
Record Dates: First submitted 2024-03-06; First posted 2024-04-04 (Actual); Last update posted 2024-04-23 (Actual); Status verified 2024-04

CONDITIONS: Mental Health Issue; Cognitive Symptom; Primary Health Care
MeSH Terms: conditions — Neurobehavioral Manifestations

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Saliva.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Case1: Individuals diagnosed with major depressive disorder (MDD)
- Case2: Individuals diagnosed with stress induced exhaustion disorder (SED)
  Interventions: Diagnostic Test: Cognitive Testing
- Control: Healthy Controls (HC) (i.e. individuals without symptoms of MDD or SED)
  Interventions: Diagnostic Test: Cognitive Testing

INTERVENTIONS:
Diagnostic Test: Cognitive Testing — Digital Cognitive Testing performed at home.
  Groups: Case2; Control

SUMMARY:
The PrimeCog study aims to describe the symptomatology and pathophysiology of stress-induced exhaustion disorder (SED) and major depressive disorder (MDD) compared to healthy controls (HC). The participants will be recruited at primary care centers, and samples of blood, saliva, and hair will be collected. Digital questionnaires covering psychosocial variables and screening instruments for the detection of depression, anxiety, etc., along with a digital cognitive test battery, will be performed at home. Subsequently, an MRI of the brain will be performed, and analysis of biomarkers for stress, inflammation, and neurodegeneration will be conducted. These procedures will be repeated after twelve and twenty-four months. The study will investigate differences in the biomarkers, neuroimaging findings, and cognitive abilities between patients with SED, MDD, and controls over time. Associations between the symptom severity of MDD/SED and psychosocial variables, cognition, MRI, and the biomarkers will also be examined. The aim is to provide new diagnostic tools for differentiation between MDD and SED and guide individualized treatment based on underlying pathophysiology and cognitive function. All necessary competences for conducting this extensive study are represented within the research group. The PrimeCog study is unique in its comprehensive design, addressing knowledge gaps, and directly comparing these diagnoses over time in primary care, where patients are typically treated.

DETAILED DESCRIPTION:
Research problems and specific questions Major depressive disorder (MDD) and stress induced exhaustion disorder (SED) are two growing public health concerns in primary care, causing individual suffering and affecting work productivity. MDD and SED call for different treatment strategies, but diagnosis differentiation pose several difficulties. Both conditions are linked to stress-related factors at work, and prescribed sick leave is a common treatment strategy. The main reasons for sick leave in DEP and UMS is cognitive difficulties, but no objective measures of cognition is used today. The aim of the PrimeCog project is to provide new diagnostic tools for differentiation between MDD and SED and guide individualized treatment based on cognitive function and underlying pathophysiology.

Data and method The project is a multicenter longitudinal, prospective research project on patients with newly diagnosed MDD or SED and healthy controls, n=100/group. The participants will be recruited at primary care centers. Data is collected through a digital cognitive test battery carried out at home, a questionnaire with screening scales and psychosocial risk factors, biomarkers in blood, saliva and hair, and a magnetic resonance imaging (MRI) of the brain. These procedures will be repeated after 12 and 24 months.

Societal relevance and utilization New diagnostic tools are needed for DEP and UMS in primary care to improve differential diagnosis and to individualize treatment in order to get the right intervention and treatment as quickly as possible. This could hypothetically contribute to shorter illness duration and reduce the length of sick leave. By investigating digital cognitive testing in primary care patients with MDD or SED, the PrimeCog project seeks to enhance diagnosis and follow-up which may prevent negative outcomes for individuals and benefit society by advancing mental health care as a whole. Digital cognitive testing is a new tool in primary care, and potentially both time- and cost-effective approach for objectively measuring cognitive symptoms.

ELIGIBILITY:
Inclusion Criteria:

1. adults 18 to 65 years old;
2. fluent in Swedish;
3. corrected to normal vision and hearing;
4. (for cases), newly diagnosed with MDD or SED (i.e., received as new diagnosis at the visit to the physician) according to the diagnostic criteria from DSM-V (MDD) and the Swedish Board of Health and Welfare (SED)

Exclusion Criteria:

1. already ongoing treatment for MDD/SED or previous diagnosis of MDD/SED within the last year;
2. history of serious mental illness (defined as mental illness that has required psychiatric in-patient care);
3. acute cerebrovascular event or severe head trauma in the last 6 months;
4. known cognitive impairment;
5. substance dependence, ongoing or past;
6. motor disability or impairment affecting interaction with the digital tests;
7. photosensitive epilepsy or -migraines.

For the MRI subgroup, any contraindication to MRI is an exclusion criterion.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients and controls in primary care.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2024-04-01 (Actual); Primary Completion 2027-04-01 (Estimated); Study Completion 2029-04-01 (Estimated)

PRIMARY OUTCOMES:
Cognitive Test Results regarding attention and processing speed | At baseline, i.e. at diagnosis, at first study-specific follow-up (12 months from baseline), and at second study-specific follow-up (24 months from baseline)
  How do cognitive test results regarding attention and processing speed measured by TMT-A vary between individuals with MDD/SED and HC?
Cognitive Test Results regarding attention and processing speed | At baseline, i.e. at diagnosis, at first study-specific follow-up (12 months from baseline), and at second study-specific follow-up (24 months from baseline)
  How do cognitive test results regarding attention and processing speed measured by TMT-B vary between individuals with MDD/SED and HC?
Cognitive Test Results regarding attention and processing speed | At baseline, i.e. at diagnosis, at first study-specific follow-up (12 months from baseline), and at second study-specific follow-up (24 months from baseline)
  How do cognitive test results regarding attention and processing speed measured by SDPTvary between individuals with MDD/SED and HC?
Cognitive Test Results regarding attention and processing speed | At baseline, i.e. at diagnosis, at first study-specific follow-up (12 months from baseline), and at second study-specific follow-up (24 months from baseline)
  How do cognitive test results regarding attention and processing speed measured by Reaction Time Test Simple vary between individuals with MDD/SED and HC?
Cognitive Test Results regarding memory | At baseline, i.e. at diagnosis, at first study-specific follow-up (12 months from baseline), and at second study-specific follow-up (24 months from baseline)
  How do cognitive test results regarding memory, measured by Corsi Span forward and backward, vary between individuals with MDD/SED and HC?
Cognitive Test Results regarding memory | At baseline, i.e. at diagnosis, at first study-specific follow-up (12 months from baseline), and at second study-specific follow-up (24 months from baseline)
  How do cognitive test results regarding memory, measured by RAVLT Learning and Recall vary between individuals with MDD/SED and HC?
Cognitive Test Results regarding executive function | At baseline, i.e. at diagnosis, at first study-specific follow-up (12 months from baseline), and at second study-specific follow-up (24 months from baseline)
  How do cognitive test results regarding executive functions, measured by TMT-B, vary between individuals with MDD/SED and HC?
Cognitive Test Results regarding executive function | At baseline, i.e. at diagnosis, at first study-specific follow-up (12 months from baseline), and at second study-specific follow-up (24 months from baseline)
  How do cognitive test results regarding executive functions, measured by Reaction Time Test Complex (or CPT) vary between individuals with MDD/SED and HC?
Cognitive Test Results regarding executive function | At baseline, i.e. at diagnosis, at first study-specific follow-up (12 months from baseline), and at second study-specific follow-up (24 months from baseline)
  How do cognitive test results regarding executive functions, measured by Stroop Test vary between individuals with MDD/SED and HC?
Cognitive Test Results regarding language | At baseline, i.e. at diagnosis, at first study-specific follow-up (12 months from baseline), and at second study-specific follow-up (24 months from baseline)
  How do cognitive test results regarding language, measured by FAS vary between individuals with MDD/SED and HC?
Cognitive Test Results regarding language | At baseline, i.e. at diagnosis, at first study-specific follow-up (12 months from baseline), and at second study-specific follow-up (24 months from baseline)
  How do cognitive test results regarding language, measured by Boston Naming Test vary between individuals with MDD/SED and HC?
Cognitive Test Results regarding visuospatial capacity | At baseline, i.e. at diagnosis, at first study-specific follow-up (12 months from baseline), and at second study-specific follow-up (24 months from baseline)
  How do cognitive test results regarding visuospatial capacity measured by: Cube Copying Test, vary between individuals with MDD/SED and HC?

SECONDARY OUTCOMES:
MRI features, measured by morphological and quantitative MR sequences of the brain | At baseline, i.e. at diagnosis, at first study-specific follow-up (12 months from baseline), and at second study-specific follow-up (24 months from baseline)
  How do morphological as well as quantitative MR sequences, with and without intravenous contrast agent with following vary between individuals with MDD/SED and HC?
Biochemical Profile in blood regarding inflammation, stress and neurodegeneration | At baseline, i.e. at diagnosis, at first study-specific follow-up (12 months from baseline), and at second study-specific follow-up (24 months from baseline)
  How the biochemical profile in blood vary between individuals with MDD/SED and HC?
Biochemical Profile in saliva regarding inflammation and stress | At baseline, i.e. at diagnosis, at first study-specific follow-up (12 months from baseline), and at second study-specific follow-up (24 months from baseline)
  How the biochemical profile in saliva as described above vary between individuals with MDD/SED and HC?
Biochemical Profile in hair regarding exposure to stress | At baseline, i.e. at diagnosis, at first study-specific follow-up (12 months from baseline), and at second study-specific follow-up (24 months from baseline)
  How the biochemical profile in hair as described above vary between individuals with MDD/SED and HC?

CONTACTS AND LOCATIONS:
Overall Officials: Hanna Israelsson Larsen, PhD, Principal Investigator — Region Ostergotland/Linkoping University; Anna Segernas, PhD, Principal Investigator — Region Ostergotland/Linkoping University
Locations (1):
- Region Ostergotland, primary care centrum, Linköping, Östergötland County, Sweden

IPD SHARING:
Plan to Share IPD: Undecided
Probably upon request from mandated researchers, but yet to be decided.